CLINICAL TRIAL: NCT04306575
Title: Challenges and Complications of a Stepwise Approach for Transvenous Lead Extraction, Single High-Volume Center Study
Brief Title: Complications of a Stepwise Approach for Transvenous Lead Extraction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Aboelhassan Abdelrady Mohamed, Assistant lecturer, Assiut University
Other Study IDs: 01020031284
Record Dates: First submitted 2020-02-29; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Pacemaker Lead Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Trans-venous lead extraction — Patients with a dysfunction or infection of a cardiac pacemaker or a defibrillator are indicated for extraction of these devices, so lead extraction is done transvenously to remove these leads

SUMMARY:
It is an observational study of predictors of complications and difficulty of trans-venous lead extraction procedure. This procedure is done for patient who had a previous cardiac pacemaker or defibrillator implantation which had a dysfunction or infection so needed to be extracted.

DETAILED DESCRIPTION:
The number of cardiac implantable electronic device (CIED) implantations has increased over recent years (1) with approximately 1.2-1.4 million CIEDs are being implanted annually worldwide.(2) Consequently this has been associated with increasing rates of infection and lead malfunctions, affecting approximately 1-2% of all CIED cases.(3)

Recently, it is estimated that between 10 000 and 15 000 leads are extracted worldwide each year.(4) Over the past few decades, transvenous lead extraction (TLE) has evolved as the preferred method for leads removal being less invasive compared to surgical removal by open heart surgery which is now reserved for cases with high risk procedures or a very large vegetation.

Most frequent indications for TLE are infection (accounting for 52.8%) and lead dysfunction (accounting for 38.1%) of all cases of TLE. (5)

There have been different approaches (superior and inferior approaches) and techniques for TLE. Current techniques employ mechanical and/or laser equipment with variable success rates. The locking stylet has been the principal tool in these techniques, while the telescoping (powered or non-powered) mechanical or laser sheaths serve as the most important ancillary tools.

Despite being a safe procedure with minor complications ranging from 0.06 to 6.2%, but serious complications may still arise in 0.2-1.8 % of cases in even the most experienced hands with mortality rates in several large registries amounting 0.2 - 1.2 %.(6) Although many studies have tried to identify risk factors for complications including patient/lead profile and centre/operator experience, major studies still have conflicting results.

Recently, the hybrid approach, with mini-thoracotomy or thoracoscopy, has been introduced and supposed to be associated with increased safety in challenging TLE procedures. (7, 8)

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients referred for lead extraction with class I and IIa indications according to 2017 HRS expert consensus statement on CIED lead management and extraction.

Exclusion Criteria:

* Patients primarily requiring surgical extraction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All ages and genders indicated for the procedure are recruited and all patient clinical background, morbidity and pacemaker related data will be collected
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Procedural related major complications | one year
  Complications includes pericardial effusion/tamponade, arrhythmia, hypotension, pulmonary embolism and death

SECONDARY OUTCOMES:
Clinical and radiological success | 3 months
  clinical success means that the procedure completed with no procedural complications, Radiological success means complete extraction of the whole lead or remaining of less than 3 cm

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curnis, Principal Investigator — Assiut University
Locations (1):
- Brescia university hospital, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Curnis A, Bontempi L, Coppola G, Cerini M, Gennaro F, Vassanelli F, Lipari A, Ashofair N, Pagnoni C, Bisleri G, Munaretto C, Dei Cas L. Active-fixation coronary sinus pacing lead extraction: a hybrid approach. Int J Cardiol. 2012 May 3;156(3):e51-2. doi: 10.1016/j.ijcard.2011.08.016. Epub 2011 Sep 9. No abstract available. PMID 21907423
- [Background] Bontempi L, Vassanelli F, Cerini M, Bisleri G, Repossini A, Giroletti L, Inama L, Salghetti F, Liberto D, Giacopelli D, Raweh A, Muneretto C, Curnis A. Hybrid Minimally Invasive Approach for Transvenous Lead Extraction: A Feasible Technique in High-Risk Patients. J Cardiovasc Electrophysiol. 2017 Apr;28(4):466-473. doi: 10.1111/jce.13164. Epub 2017 Feb 9. PMID 28063271